CLINICAL TRIAL: NCT00904488
Title: Addition of Oral Metolazone to Intermittent Intravenous Furosemide Versus Transition to Continuous Infusion Furosemide in Acute Decompensated Heart Failure Patients Experiencing an Inadequate Response to Therapy
Brief Title: Oral Metolazone and Intermittent Intravenous Furosemide Versus Continuous Infusion Furosemide in Acute Heart Failure
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficult recruitment
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: University of Illinois at Chicago (Other); Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-1292
Record Dates: First submitted 2009-05-17; First posted 2009-05-19 (Estimated); Results first posted 2018-02-13 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-01

CONDITIONS: Acute Decompensated Heart Failure
Keywords: Acute Decompensated Heart Failure; Diuretics
MeSH Terms: interventions — Metolazone; Furosemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Addition of PO Thiazide Diuretic (Active Comparator): Addition of oral metolazone 5 mg daily to current intravenous bolus furosemide. All subjects will continue their current dose of intravenous bolus furosemide.
  Interventions: Drug: Addition of oral Metolazone
- IV furosemide dose escalation (Active Comparator): Current IV furosemide dose will be escalated to 2-2.5 x current dose, given as either IV bolus or continuous infusion over 24 hours.
  Interventions: Drug: Furosemide dose escalation

INTERVENTIONS:
Drug: Addition of oral Metolazone — Addition of oral metolazone 5 mg daily to continued current dose of intravenous bolus furosemide
  Other Names: Zaroxolyn
  Arms: Addition of PO Thiazide Diuretic
Drug: Furosemide dose escalation — Furosemide dose escalation via either IV bolus (2-2.5 x current dose) or continuous infusion (2-2.5 x current dose administered over previous 24 hours)
  Other Names: Lasix
  Arms: IV furosemide dose escalation

SUMMARY:
The purpose of this prospective, randomized, open-label study is to compare two diuretic strategies in patients with acute decompensated heart failure (ADHF): the addition of an oral thiazide diuretic to intravenous bolus (IVB) loop diuretic will be compared to transition from IVB to continuous infusion (CI) loop diuretic.

DETAILED DESCRIPTION:
Patients hospitalized for ADHF secondary to fluid overload and who are experiencing an inadequate response to IVB furosemide and require additional diuresis will be enrolled. Patients will be randomized to one of two treatment arms: the addition of oral metolazone to continued IVB furosemide versus transition from IVB to CI furosemide. A suggested algorithm for initial dosing and titration of these two diuretic strategies will be provided. Baseline and daily data collection will include various efficacy and safety endpoints including daily net urine output and weight, patient and physician global assessment scale, length of stay, 30-day death or rehospitalization, vital signs, electrolytes, and renal function. Clinically meaningful efficacy and safety endpoints will be compared.

ELIGIBILITY:
Inclusion Criteria:

1. Greater than or equal to 18 years of age
2. Hospitalized for acute decompensated heart failure (ADHF) secondary to fluid overload as defined by the presence of at least

   * 1 symptom (e.g. dyspnea, orthopnea, paroxysmal nocturnal dyspnea) AND
   * 1 sign (e.g. rales on auscultation, > 2+ peripheral or presacral> edema, hepatomegaly, ascites, jugular vein distension > 7 cm, pulmonary vascular congestion on chest radiography)
3. Inadequate response to IV diuretics and requiring additional diuresis as determined by primary medical team
4. Received less than six doses of IV furosemide OR enrolled within 72 hours of hospital admission
5. Anticipated need for intravenous diuretic therapy for at least 48 hours
6. Able to provide informed consent

Exclusion Criteria:

1. Receiving a continuous infusion loop diuretic during current hospital visit
2. Substantial diuretic response to pre-randomization diuretic dosing such that higher doses of diuretic would be contraindicated (based on judgement of patient's primary team)
3. Planned or ongoing intravenous vasoactive therapy (e.g. inotrope, vasodilator) or mechanical support (e.g. intra-aortic balloon pump, ventricular assist device) for ADHF during this hospitalization
4. Planned elective admission for elective placement/revision of a cardiovascular device (e.g. defibrillator, biventricular pacemaker) during this hospitalization or such within the preceding 7 days
5. Systolic blood pressure < 90 mmHg
6. Serum creatinine > 3 mg/dL at baseline or renal replacement therapy including ultrafiltration
7. Serum potassium < 3.5 mEq/L (3.0 - 3.4 mEq/L allowed if supplemental potassium is being administered)
8. Serum magnesium < 1.6 mg/dL (1.4 - 1.5 mg/dL allowed if supplemental magnesium is being administered)
9. Acute coronary syndrome or hemodynamically significant arrhythmias causing worsening HF
10. Severe, uncorrected primary cardiac valvular disease, acute myocarditis, constrictive pericarditis, hypertrophic obstructive cardiomyopathy, restrictive or constrictive cardiomyopathy, complex congenital heart disease
11. Primary pulmonary hypertension with right sided heart failure
12. Use of iodinated radiocontrast material in prior 72 hours or planned within the next 48 hours
13. Enrollment or planned enrollment in another randomized clinical trial during hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-10 (Actual); Primary Completion 2016-05-28 (Actual); Study Completion 2017-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jo E. Rodgers, PharmD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC_Chapel Hill, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Furosemide Dose Escalation: Furosemide dose escalation given either as IV bolus (2-2.5 x current dose) or continuous infusion (2-2.5 x current dose administered over previous 24 hours)
- IVB Loop and PO Thiazide Diuretic: Addition of oral metolazone 5 mg daily to continued intravenous bolus furosemide (Furosemide continued at current dose)
Period: Overall Study
Arm/Group | Furosemide Dose Escalation | IVB Loop and PO Thiazide Diuretic
Started | 5 | 6
Completed | 5 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Furosemide Dose Escalation: IV furosemide dose escalation via either intravenous bolus (2-2.5 x current dose) or continuous infusion furosemide (Furosemide 2-2.5 x current dose administered over previous 24 hours)
- Total: Total of all reporting groups
Arm/Group | Furosemide Dose Escalation | IVB Loop and PO Thiazide Diuretic | Total
Number analyzed (Participants) | 5 | 6 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (16.0) | 55.8 (16.2) | 56.6 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 2 | 4 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 2 | 3 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 6 | 11
Baseline Ejection Fraction (EF) (%) [Count of Participants; unit: Participants]
  Mild (55-60%) | 2 | 1 | 3
  Moderate (20-40%) | 1 | 5 | 6
  Severe (5-15%) | 2 | 0 | 2
Chief Complaints [Number; unit: participants]
  Shortness of Breath (SOB) | 2 | 2 | 3
  Weight Gain | 0 | 1 | 1
  Fluid Overload | 1 | 2 | 2
Afib on Admission [Count of Participants; unit: Participants]
  Present | 0 | 0 | 0
  Absent | 3 | 5 | 8
  Not reported | 2 | 1 | 3
New York Heart Association (NYHA) Class on Admission [Count of Participants; unit: Participants] — ClassI No limitation of physical activity. Best outcome.
  ClassII Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea (shortness of breath).
  ClassIII Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea.
  ClassIV Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest. If any physical activity is undertaken, discomfort increases. Worst outcome
  Participants
    Class I | 0 | 0 | 0
    Class II | 0 | 0 | 0
    Class III | 0 | 3 | 3
    Class IV | 1 | 1 | 2
    Not Reported | 4 | 2 | 6
Comorbidities [Number; unit: participants]
  Anemia | 2 | 0 | 2
  Coronary artery disease (CAD) | 1 | 3 | 4
  Chronic obstructive pulmonary disease (COPD) | 0 | 2 | 2
  Cerebrovascular accident (CVA) | 1 | 2 | 3
  Diabetes | 4 | 3 | 7
  Dyslipidemia | 4 | 2 | 6
  Gastroesophageal reflux disease (GERD) | 1 | 0 | 1
  Gout | 1 | 1 | 2
  Human immunodeficiency virus (HIV) | 1 | 0 | 1
  Myocardial infarction (MI) | 1 | 1 | 2
  Hypertension | 4 | 4 | 8
  Obesity | 2 | 1 | 3
  Obstructive Sleep Apnea | 2 | 2 | 4
Medication [Number; unit: participants]
  Beta Blocker | 4 | 4 | 8
  Angiotensin-converting-enzyme inhibitor | 4 | 6 | 10
  Angiotensin Receptor Blockers | 0 | 0 | 0
  Loop Diuretic | 4 | 5 | 9
  Aldosterone Antagonist | 0 | 1 | 1
  Digoxin | 2 | 0 | 2
  Calcium Channel Blocker | 2 | 1 | 3
  Isosorbide Dinitrate | 1 | 1 | 2
  Hydralazine | 4 | 1 | 5
  Statin | 5 | 4 | 9
  Anticoagulant | 2 | 3 | 5
  Aspirin | 2 | 5 | 7
  Potassium supplement | 1 | 3 | 4
Brain Natriuretic Peptide (BNP) at admission [Mean (Standard Deviation); unit: pg/ml] — Population: BNP was not measured on admission as part of routine clinical care in all subjects.
  pg/ml
    number analyzed (Participants) | 4 | 3 | 7
    (all) | 6800.75 (10330.95) | 5401.33 (4183.06) | 6201.00 (7313.54)

OUTCOME MEASURES:

1. Primary Outcome: Daily Net Fluid Output on Day 2 (24-48 Hours After Randomization)
Description: Net fluid output = fluid output during 24-48 hours after randomization - fluid intake during 24-48 hours after randomization. A negative value means that daily fluid intake was less than the daily fluid output.
Time Frame: 24-48 hours
Measure: Mean (Standard Deviation); unit: mL/day
Arm/Group | Furosemide Dose Escalation | IVB Loop and PO Thiazide Diuretic
Number analyzed (Participants) | 5 | 6
mL/day | -1454.60 (1339.53) | -1322.83 (1738.30)

2. Secondary Outcome: Daily Net Fluid Output on Days 1, 3, and 4
Description: Daily net fluid output = daily fluid output - daily intake. A negative value means that daily fluid intake was less than the daily fluid output.
Time Frame: 0-24, 48-72, 72-96 hrs
Population: If diuretic therapy is changed to the oral route before a scheduled efficacy endpoint is to be measured (e.g.72 or 96 hour net output), then that endpoint will not be obtained.
Measure: Mean (Standard Deviation); unit: ml/day
Arm/Group | Furosemide Dose Escalation | IVB Loop and PO Thiazide Diuretic
Number analyzed (Participants) | 5 | 6
ml/day
  0-24 hr | -2226.74 (2063.63) | -3076.67 (1555.63)
  48-72 hr: number analyzed (Participants) | 4 | 5
  48-72 hr | -2108.00 (2187.05) | -409.74 (1208.98)
  72-96 hr: number analyzed (Participants) | 3 | 3
  72-96 hr | -2433.33 (1374.38) | -705.33 (157.39)

3. Secondary Outcome: Daily Urine Output (mL Urine Out Per mg Furosemide (IV Equivalent) Received)
Time Frame: 0-24, 24-48, 48-72, 72-96 hrs
Population: Data were not collected at all time points for all subjects, and were only analyzed when available. Data not analyzed on days when diuretics were held or discontinued.
Measure: Mean (Standard Deviation); unit: ml/mg furosemide received
Arm/Group | Furosemide Dose Escalation | IVB Loop and PO Thiazide Diuretic
Number analyzed (Participants) | 5 | 6
ml/mg furosemide received
  0-24 hr | 29.35 (21.01) | 17.35 (7.11)
  24-48 hr: number analyzed (Participants) | 2 | 5
  24-48 hr | 8.28 (4.59) | 21.88 (14.39)
  48-72 hr: number analyzed (Participants) | 4 | 3
  48-72 hr | 25.84 (20.05) | 25.52 (14.84)
  72-96 hr: number analyzed (Participants) | 2 | 0
  72-96 hr | 43.94 (28.12) |

4. Secondary Outcome: Daily Weight
Time Frame: Baseline (Dry), Baseline, 0-24, 24-48, 48-72, 72-96 hrs
Population: Data were not collected for all subjects at all time points, and were only analyzed when available
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Furosemide Dose Escalation | IVB Loop and PO Thiazide Diuretic
Number analyzed (Participants) | 5 | 6
Kg
  Baseline (Dry): number analyzed (Participants) | 4 | 5
  Baseline (Dry) | 82.35 (40.87) | 100.82 (49.35)
  Baseline | 120.84 (75.25) | 102.57 (33.57)
  0-24 hr: number analyzed (Participants) | 3 | 6
  0-24 hr | 154.23 (103.30) | 101.07 (32.88)
  24-48 hr: number analyzed (Participants) | 4 | 6
  24-48 hr | 129.73 (91.46) | 99.08 (32.93)
  48-72 hr: number analyzed (Participants) | 3 | 5
  48-72 hr | 135.07 (101.31) | 106.70 (52.18)
  72-96 hr: number analyzed (Participants) | 2 | 3
  72-96 hr | 172.10 (107.71) | 86.87 (48.17)

5. Secondary Outcome: Patient Global Assessment Scale
Description: Scale range: 1-5 Which of the following best describes your overall health state today?
  1. = markedly worse
  2. = worse
  3. = neither better nor worse
  4. = better
  5. = markedly better
Time Frame: Baseline, 24, 48, 72, 96 hrs
Population: Data were not collected at all time points, and were only analyzed when available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Furosemide Dose Escalation | IVB Loop and PO Thiazide Diuretic
Number analyzed (Participants) | 5 | 6
units on a scale
  Baseline: number analyzed (Participants) | 4 | 3
  Baseline | 3.25 (1.67) | 3.67 (2.23)
  24 hr: number analyzed (Participants) | 5 | 4
  24 hr | 4.2 (0.45) | 4.25 (2.23)
  48 hr: number analyzed (Participants) | 5 | 5
  48 hr | 3.8 (1.1) | 3.6 (1.67)
  72 hr: number analyzed (Participants) | 3 | 4
  72 hr | 4.67 (2.59) | 3.75 (1.97)
  96 hr: number analyzed (Participants) | 2 | 3
  96 hr | 4 (2.19) | 4 (2.19)

6. Secondary Outcome: Physician Global Assessment Scale
Description: Scale range: 1-5 Which of the following best describes the patient's overall health state today?
  1. = markedly worse
  2. = worse
  3. = neither better nor worse
  4. = better
  5. = markedly better
Time Frame: Baseline, 24, 48, 72, 96 hours
Population: Data were not collected at all time points, and were only analyzed when available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Furosemide Dose Escalation | IVB Loop and PO Thiazide Diuretic
Number analyzed (Participants) | 5 | 6
units on a scale
  Baseline: number analyzed (Participants) | 3 | 2
  Baseline | 2.67 (1.67) | 2 (1.21)
  24 hr: number analyzed (Participants) | 4 | 4
  24 hr | 4.25 (1.95) | 4 (2.16)
  48 hr: number analyzed (Participants) | 4 | 5
  48 hr | 4 (1.92) | 4 (1.63)
  72 hr: number analyzed (Participants) | 2 | 4
  72 hr | 4.5 (2.49) | 3.75 (1.97)
  96 hr: number analyzed (Participants) | 2 | 4
  96 hr | 4 (2.19) | 3.67 (2.19)

7. Secondary Outcome: Need for Additional or Alternative Diuretic (Crossover) or Other Vasoactive Therapy (Study Failure)
Description: Patients will be considered a treatment failure if they require additional diuretic (including crossover to the alternative study arm) or require IV vasoactive drug therapy (e.g. vasodilators including nitroglycerin or inotropes) as deemed appropriate/necessary by their medical team.
Time Frame: 0-96 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Furosemide Dose Escalation | IVB Loop and PO Thiazide Diuretic
Number analyzed (Participants) | 5 | 6
Participants | 1 | 4

8. Secondary Outcome: Time to Return to Baseline Weight
Time Frame: 0-96 hours
Population: Weight was not collected in all subjects every day.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Furosemide Dose Escalation | IVB Loop and PO Thiazide Diuretic
Number analyzed (Participants) | 4 | 6
Days | 1.5 (1.1) | 1.5 (0.84)

9. Secondary Outcome: Length of Hospitalization
Time Frame: Assessed till hospital discharge, an average of 1 week (longest 29 days)
Population: Data not available in all subjects.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Furosemide Dose Escalation | IVB Loop and PO Thiazide Diuretic
Number analyzed (Participants) | 4 | 4
Days | 4.75 (1.71) | 11.25 (10.93)

10. Secondary Outcome: 30-day All-cause Mortality
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Furosemide Dose Escalation | IVB Loop and PO Thiazide Diuretic
Number analyzed (Participants) | 5 | 6
Participants | 0 | 0

11. Secondary Outcome: Rehospitalization at 30 Days
Time Frame: 30 days
Population: 30-day follow up data (except for mortality) were not collected in 2 participants
Measure: Count of Participants; unit: Participants
Arm/Group | Furosemide Dose Escalation | IVB Loop and PO Thiazide Diuretic
Number analyzed (Participants) | 4 | 5
Participants | 1 | 1

12. Secondary Outcome: Unscheduled Heart Failure Visits to Emergency Department or Outpatient Clinic
Time Frame: 30 days
Population: 30-day follow up data (except for mortality) were not collected in 2 participants
Measure: Count of Participants; unit: Participants
Arm/Group | Furosemide Dose Escalation | IVB Loop and PO Thiazide Diuretic
Number analyzed (Participants) | 4 | 5
Participants | 1 | 1

13. Secondary Outcome: Blood Urea Nitrogen (BUN)
Time Frame: Baseline, 24, 48, 72, 96 hours
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Furosemide Dose Escalation | IVB Loop and PO Thiazide Diuretic
Number analyzed (Participants) | 5 | 6
mg/dL
  Baseline | 31.20 (11.05) | 29.83 (16.82)
  24 hr | 28.00 (9.35) | 27.67 (17.18)
  48 hr | 30.80 (11.45) | 33.17 (16.92)
  72 hr | 29.00 (12.08) | 42.00 (20.70)
  96 hr | 38.60 (19.63) | 42.67 (20.63)

ADVERSE EVENTS:
Time Frame: Changes in labs and vitals were collected for 96 hours after randomization All-cause mortality were collected for 30 days after randomization
Description: * Total number of times antihypertensive doses are held due to low blood pressure
  * Number of hypotensive episodes defined as systolic blood pressure below 85 mmHg or greater than 10 mmHg below baseline (whichever is greater)
  * Number of critically low potassium (< 3.5 mmol/L) and magnesium (< 1.6 mg/dL) concentrations while receiving study therapy
Arm/Group | Furosemide Dose Escalation | IVB Loop and PO Thiazide Diuretic
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 2/5 | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Furosemide Dose Escalation (N=5) | IVB Loop and PO Thiazide Diuretic (N=6)
critically low potassium (< 3.5 mmol/L) while receiving study therapy (Cardiac disorders) | 0 (0) | 1 (1)
critically low magnesium (< 1.6 mg/dL) while receiving study therapy (Cardiac disorders) | 0 (0) | 1 (1)
Hypotension (Cardiac disorders) | 2 (8) | 6 (32)
Hypotension resulting in holding antihypertensive doses (Cardiac disorders) | 0 (0) | 1 (8) — Reported as number of subjects affected/total at risk. Count of occurrence is total number of doses of antihypertensives being held.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes